CLINICAL TRIAL: NCT00748228
Title: Dopamine in Orthostatic Tolerance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is being replaced by another protocol.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Emily M. Garland, Research Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 040769; HL071784
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Postural Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Sodium, Dietary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): 10 mEq/day dietary sodium
  Interventions: Dietary Supplement: dietary sodium
- B (Experimental): 150 mEq/day dietary sodium
  Interventions: Dietary Supplement: dietary sodium
- C (Experimental): 300 mEq/day dietary sodium
  Interventions: Dietary Supplement: dietary sodium

INTERVENTIONS:
Dietary Supplement: dietary sodium — 10 mEq/day
  Arms: A
Dietary Supplement: dietary sodium — 300 mEq/day
  Arms: C
Dietary Supplement: dietary sodium — 150 mEq/day dietary sodium
  Arms: B

SUMMARY:
One goal of this study is to determine whether people with different amounts of dopamine-beta-hydroxylase (DBH) have different responses to events that affect blood pressure and heart rate. We will also study whether increasing dietary salt improves symptoms during upright posture. Finally, we will examine whether the dietary sodium level influences serum DBH activity and whether DBH level influences the response to sodium. DBH levels and the function of the sympathetic or involuntary nervous system will be assessed in normal volunteers and in patients with postural tachycardia syndrome (POTS).

ELIGIBILITY:
Inclusion Criteria:

* Upright plasma norepinephrine > 600 pg/ml, or
* An increase in heart rate of > 30 beats per minute upon standing, and
* Withdrawal of all medications for at least 3 days, and
* No associated medical illness, and
* Age 18 - 60 years old.

Exclusion Criteria:

* Older than 60 years of age
* Routinely taking medications affecting the autonomic nervous system
* Any chronic illness (cardiac, pulmonary, endocrine, gastrointestinal, rheumatologic) other than POTS
* Anemia (Hct < 30)
* Women of childbearing age who are pregnant or nursing
* Unable to give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2004-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
plasma dopamine-beta-hydroxylase | at enrollment and after tests
plasma dopamine | after tests

CONTACTS AND LOCATIONS:
Overall Officials: Emily M Garland, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States